CLINICAL TRIAL: NCT00005022
Title: A Phase I/II Escalation Study of Thoracic Irradiation With Concurrent Chemotherapy for Patients With Limited Small Cell Lung Cancer
Brief Title: Radiation Therapy Plus Combination Chemotherapy in Treating Patients With Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-9712; CDR0000065797
Record Dates: First submitted 2000-04-06; First posted 2004-01-29 (Estimated); Last update posted 2013-11-04 (Estimated); Status verified 2013-10

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Cisplatin; Etoposide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Arm 1 (Experimental): Large field radiation therapy 36 Gy, 1.8 Gy/fx/D/5 days/4 weeks, boost 1.8 Gy/D x 2 days, then BID x last 3 days.
  Interventions: Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy
- Arm 2 (Experimental): Large field radiation therapy 36 Gy, 1.8 Gy/fx/D/5 days/4 weeks, boost 1.8 Gy/BID x last 5 days.
  Interventions: Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy
- Arm 3 (Experimental): Large field radiation therapy 32.4 Gy, 1.8 Gy/fx/D/5 days x 18 fx, boost just in pm @ 1.8 Gy/fx on days 19 & 20, then boost 1.8 Gy BID x last 5 days.
  Interventions: Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy
- Arm 4 (Experimental): Large field radiation therapy 28.8 Gy, 1.8 Gy/fx/5 days x 16 fx, boost just in pm @ 1.8 Gy/fx on days 17-20, then boost 1.8 Gy BID x last 5 days.
  Interventions: Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy
- Arm 5 (Experimental): Large field radiation therapy 36 Gy, 1.8 Gy/fx/D 5 days/4 weeks, boost 1.8 Gy/D x 2 days, then BID x last 3 days.
  Interventions: Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy
- Arm 6 (Experimental): Large field radiation therapy 25.2 Gy, 1.8 Gy/fx/5 days x 14 fx, boost just in pm @ 1.8 Gy/fx on days 15-20, then boost 1.8 Gy BID x last 5 days.
  Interventions: Drug: cisplatin; Drug: etoposide; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: etoposide
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one chemotherapy drug with radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of radiation therapy plus combination chemotherapy in treating patients with limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of thoracic radiation using an accelerated boost with concurrent chemotherapy in patients with small cell lung cancer. II. Evaluate the response rate and overall survival in these patients. III. Reduce the toxic effects of treatment to esophagus and lungs.

OUTLINE: This is a radiation dose escalation study. Patients are sequentially accrued to one of four radiation dose levels. Dose level 1: Patients receive radiotherapy 5 days a week for 4 weeks followed by radiation boost given daily for 2 days, then twice daily for 3 days during week 5. (Closed to accrual 6/98) Dose level 2: Patients receive radiotherapy 5 days a week for 4 weeks followed by radiation boost given twice daily for 5 days during week 5. (Closed to accrual 9/24/99) Dose level 3: Patients receive radiotherapy 5 days a week for 18 days followed by radiation boost given in the evenings on days 19 and 20, then twice daily for 5 days during week 5. (Closed to accrual 5/5/00) Dose level 4: Patients receive radiotherapy 5 days a week for 16 days followed by radiation boost given in the evenings on days 17-20, then twice daily for 5 days during week 5. The fifth dose level is the same as the first dose level. (Closed to accrual 3/19/99) Cohorts of 5 patients are entered at each radiation dose level. If one patient experiences nonhematologic dose limiting toxicity (DLT), 5 additional patients are treated at that level. If no further DLT occurs, escalation to the next arm proceeds. Patients receive cisplatin IV plus etoposide IV on day 1 of radiotherapy and oral etoposide on days 2 and 3 every 3 weeks for 4 courses. Patients are followed every 3 months for 1 year, every 6 months for 2 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study within 5-10 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed small cell carcinoma of the lung Limited disease (stage I-IIIb but excluding T4 tumor based on malignant pleural effusion or N3 disease based on contralateral hilar or contralateral supraclavicular involvement) No pericardial or pleural effusion on chest x-ray regardless of cytology Measurable or evaluable disease Tumor must be encompassed by limited radiation therapy fields without causing severe symptomatic pulmonary dysfunction

PATIENT CHARACTERISTICS: Age: 18 to 80 Performance status: Karnofsky 70-100% Life expectancy: Greater than 6 months Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 150,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Cardiovascular: No symptomatic heart disease At least 6 months since prior myocardial infarction Pulmonary: See Disease Characteristics Forced expiratory volume at one second (FEV1) greater than 0.8 L No uncontrolled bronchospasm in unaffected lung Other: No other serious concurrent illness No prior or concurrent malignancy within the past 2 years except curatively treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No other concurrent malignancy No history of uncontrolled psychiatric illness, severe head injury, chronic alcohol or drug abuse, or central nervous system disease Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: No prior complete tumor resection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 1998-02; Primary Completion 2002-10 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Frequency of patients developing unacceptable (grade 3 or higher) acute toxicities attributable to thoracic irradiation with concurrent chemotherapy | From start of treatment until 90 days

SECONDARY OUTCOMES:
Compare baseline and follow-up Mini Mental Status Examinations | From baseline until end of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Ritsuko U. Komaki, MD, FACR, Study Chair — M.D. Anderson Cancer Center
Locations (262):
- United States (242):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Huntsville Hospital System, Huntsville, Alabama
  - Comprehensive Cancer Institute of Huntsville, Huntsville, Alabama
  - MBCCOP - Gulf Coast, Mobile, Alabama
  - Alabama Oncology, LLC, Montgomery, Alabama
  - Radiation Oncology Associates of West Alabama, Tuscallosa, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Foundation for Cancer Research and Education, Phoenix, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Mount Diablo Medical Center, Concord, California
  - Cancer Center and Beckman Research Institute, City of Hope, Duarte, California
  - California Cancer Center, Fresno, California
  - Saint Agnes Cancer Center, Fresno, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Sutter Health West Cancer Research Group, Greenbrae, California
  - University of California San Diego Cancer Center, La Jolla, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Huntington Cancer Center, Pasadena, California
  - Cancer Care Center, Pomona, California
  - Radiation Oncology Center - Sacramento, Sacramento, California
  - Radiation Medical Group, Inc., San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - O'Connor Hospital, San Jose, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Memorial Hospital Cancer Center, Colorado Springs, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - Saint Mary's Hospital and Medical Center, Grand Junction, Colorado
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Lykes Center for Radiation Therapy, Clearwater, Florida
  - Halifax Medical Center, Daytona Beach, Florida
  - Radiation Therapy Associates - Fort Myers, Fort Myers, Florida
  - University of Florida Health Science Center, Gainesville, Florida
  - Health First Holmes Regional Medical Center, Melbourne, Florida
  - Veterans Affairs Medical Center - Miami, Miami, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Florida Radiation Oncology Group, Orange Park, Florida
  - MD Anderson Cancer Center Orlando, Orlando, Florida
  - Bay Medical Center, Panama City, Florida
  - Gulf Coast Cancer Treatment Center, Panama City, Florida
  - Sarasota Radiation and Medical Oncology Center, Sarasota, Florida
  - Tallahassee Memorial Healthcare, Tallahassee, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical Center/John B. Amos Community Cancer Center, Columbus, Georgia
  - InterCommunity Cancer Center at Rome, Rome, Georgia
  - MBCCOP - Hawaii, Honolulu, Hawaii
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - CCOP - Central Illinois, Decatur, Illinois
  - Provena St. Joseph Hospital- Regional Cancer Care Center, Elgin, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - St. John's Medical Center, Anderson, Indiana
  - Bloomington Hospital, Bloomington, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - Clarion Health Partners Inc., Indianapolis, Indiana
  - Community Hospitals of Indianapolis - Regional Cancer Center, Indianapolis, Indiana
  - Ball Memorial Hospital, Muncie, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Wendt Regional Cancer Center of Finley Hospital, Dubuque, Iowa
  - Holden Comprehensive Cancer Center at The University of Iowa, Iowa City, Iowa
  - Central Baptist Hospital, Lexington, Kentucky
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - James Graham Brown Cancer Center, Louisville, Kentucky
  - Louisville Radiation Oncology, Louisville, Kentucky
  - Merle M. Mahr Cancer Center, Madisonville, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Romagosa Radiation Oncology Center, Lafayette, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Maine Medical Center, Portland, Maine
  - Anne Arundel Oncology Center, Annapolis, Maryland
  - Greater Baltimore Medical Center and Cancer Center, Baltimore, Maryland
  - Harbor Hospital Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Radiation Oncology Affiliates of Maryland, P.A., Baltimore, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Regional Cancer Center, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - MidMichigan Medical Center - Midland, Midland, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - St. Mary's Medical Center, Saginaw, Michigan
  - William Beaumont Hospital - Troy, Troy, Michigan
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - North Mississippi Medical Center/Cancer Center, Tupelo, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - Mallinckrodt Institute of Radiology, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Nebraska Health System, Omaha, Nebraska
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Elliot Regional Cancer Center, Manchester, New Hampshire
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - John F. Kennedy Medical Center, Edison, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Atlantic City Medical Center, Pomona, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Associated Radiologists, P.A., Warren Township, New Jersey
  - Saint Joseph Medical Center, Albuquerque, New Mexico
  - Cancer Center of Albany Medical Center, Albany, New York
  - State University of New York Health Science Center at Brooklyn, Brooklyn, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Finger Lakes Radiation Oncology, P.C., Clifton Springs, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Champlain Valley Physicians Hospital Medical Center, Plattsburgh, New York
  - Vassar Brothers Hospital, Poughkeepsie, New York
  - University of Rochester Cancer Center, Rochester, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Albert Einstein Comprehensive Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Riverhill Radiation Oncology, Yonkers, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Northeast Medical Center, Concord, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - Catawba Memorial Hospital, Hickory, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Meritcare Roger Maris Cancer Center, Fargo, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Akron City Hospital, Akron, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - St. Anthony Hospital, Oklahoma City, Oklahoma
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - St. John Health System, Tulsa, Oklahoma
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Hospital Regional Cancer Center, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fitzgerald Mercy Hospital, Darby, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pocono Cancer Center, East Stroudsburg, Pennsylvania
  - Penn State Geisinger Cancer Center, Hershey, Pennsylvania
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Veterans Affairs Medical Center - Philadelphia, Philadelphia, Pennsylvania
  - Kimmel Cancer Center of Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Roger Williams Medical Center/BUSM, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Jackson-Madison County General Hospital, Jackson, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Harrington Cancer Center, Amarillo, Texas
  - Julie and Ben Rogers Cancer Institute, Beaumont, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Wilford Hall - 59th Medical Wing, Lackland Air Force Base, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - East Texas Medical Center - Cancer Institute, Tyler, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center, St. George, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Green Mountain Oncology Group, Rutland, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - Cancer Center at the University of Virginia, Charlottesville, Virginia
  - RMH Regional Canter Center, Harrisonburg, Virginia
  - Naval Medical Center, Portsmouth, Portsmouth, Virginia
  - Bon-Secours - St. Mary's Hospital, Richmond, Virginia
  - Massey Cancer Center, Richmond, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Deaconess Medical Center, Spokane, Washington
  - Yakima Valley Memorial Hospital, Yakima, Washington
  - Schiffler Cancer Center, Wheeling, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Foundation, La Crosse, Wisconsin
  - Southern Wisconsin Radiotherapy Center, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Community Memorial Hospital, Menomonee Falls, Wisconsin
  - St. Joseph's Hospital, Milwaukee, Wisconsin
  - Columbia Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
  - Southeastern Wisconsin Regional Cancer Center, Racine, Wisconsin
  - Waukesha Memorial Hospital, Waukesha, Wisconsin
- Canada (20):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Newfoundland Cancer Treatment and Research Foundation, St. John's, Newfoundland and Labrador
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Northeastern Ontario Regional Cancer Centre, Sudbury, Greater Sudbury, Ontario
  - Cancer Care Ontario-Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Northwestern Ontario Regional Cancer Centre, Thunder Bay, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - CHU de Quebec - L'Hotel-Dieu de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

REFERENCES:
- [Result] Komaki R, Swann RS, Ettinger DS, Glisson BS, Sandler AB, Movsas B, Suh J, Byhardt RW. Phase I study of thoracic radiation dose escalation with concurrent chemotherapy for patients with limited small-cell lung cancer: Report of Radiation Therapy Oncology Group (RTOG) protocol 97-12. Int J Radiat Oncol Biol Phys. 2005 Jun 1;62(2):342-50. doi: 10.1016/j.ijrobp.2004.11.030. PMID 15890573
- [Result] Komaki R, Swann S, Ettinger D, et al.: Phase I dose-escalation study of thoracic irradiation with concurrent chemotherapy for patients with limited small cell lung cancer (LSCLC). Radiation Therapy Oncology Group (RTOG) protocol 9712. [Abstract] Proceedings of the American Society of Clinical Oncology 22: A-2539, 2003.